CLINICAL TRIAL: NCT05506748
Title: Association Between Preoperative HALP and Immediate Postoperative Outcomes in Patients Undergoing Pancreaticoduodenectomy
Brief Title: Association Between Preoperative HALP and Immediate Postoperative Outcomes
Status: Completed | Type: Observational
Sponsor: Chitwan Medical College (Other)
Responsible Party: Principal Investigator, Gaurav Katwal, Principal Investigator, Chitwan Medical College
Other Study IDs: 078/079-103
Record Dates: First submitted 2022-08-12; First posted 2022-08-18 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Hemoglobins; Albumins; Platelets; Lymphocytes; Morbidity; Mortality; Whipples Procedure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: pantients undergoing pancreaticoduodenectomy — The study includes all the cases who underwent pancreaticoduodenectomy for carcinoma head of the pancreas, distal cholangiocarcinoma, periampullary and duodenal cancer.

SUMMARY:
Multiple inflammation-based prognostic scores have been developed for the prediction of perioperative morbidity and mortality following pancreaticoduodenectomy (PD). Preoperative "Hemoglobin, Albumin, Lymphocytes and Platelets index (HALP)" is one of the promising inflammatory markers that has emerged as a predictor of postoperative survival. To date, no study has been done with preoperative HALP to predict 30days morbidity and mortality.

Is there any association between Preoperative HALP (hemoglobin, albumin, lymphocyte, and platelet) and 30 days post operative morbidity and mortality in patients undergoing Pancreaticoduodenectomy?

DETAILED DESCRIPTION:
General Objective:

To assess the association between preoperative HALP and immediate postoperative outcome among patients undergoing PD.

Specific Objectives:

1. To identify the magnitude of immediate post-operative morbidity and mortality in patients undergoing PD.
2. To evaluate the descriptive measurement of preoperative Hemoglobin, Albumin, Lymphocytes, Platelets and HALP among patients undergoing PD.
3. To compare the preoperative HALP with morbidity and mortality among patients undergoing PD.

Operational Definition:

1. Immediate postoperative time - was taken as 30days following surgery.
2. Morbidity- was defined by Clavién-Dindo20 grading for the surgical complication and DGE,21 POPF,22 and PPH23 -according to International Study Group of Pancreatic Surgery (ISGPS) grading.
3. Mortality- survival within 30days.
4. Level of preoperative HALP- normality test was done via SPSS and data of HALP followed normal Gaussian distribution. So, mean was used for the calculation of cut off value as 35.83. And, patients were divided into low HALP (≤35.83) group and high HALP (>35.83) group respectively

ELIGIBILITY:
Inclusion Criteria:

1. All the cases of elective pancreaticoduodenectomies for malignant pancreatic head disease

Exclusion Criteria:

1. Incomplete clinicopathological and follow-up data,
2. Age <15 years and age >80 years
3. History of antitumor treatments, and
4. Record of other malignant tumors, (unresectable?)

Ages: 15 Years to 80 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All the cases of elective pancreaticoduodenectomy with combined "Artery First with Posterior and Uncinate approach" for malignant pancreatic head disease (ampullary, HOP, dCCA, duodenal In the Department of Surgery at BPKMCH between April 2021 to April 2022.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
Morbidity- Clavién-Dindo grading : | 30days following the pancreaticoduodenectomy
  It is graded from grade I to V on the basis of surgical site infection, organ space infection, single or multiple organ failure, and death.
  Grade I Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic, and radiological interventions
  Grade II Requires pharmacological treatment, blood transfusions, or total parenteral nutrition
  Grade III Requires surgical, endoscopic, or radiological intervention IIIa Not under general anesthesia IIIb Under general anesthesia
  Grade IV Life-threatening complication requiring IC/ICU management IVa Single organ dysfunction IVb Multiorgan dysfunction
  Grade V Death of a patient
  PS- Higher the score worst the outcome.
Morbidity- Delayed Gastric Empty (DGE) | 30days following the pancreaticoduodenectomy
  Postoperative gastroparesis.
  Grade A DGE: If the Naso-Gastric Tube (NGT) is needed between the postoperative day (POD) -4 and 7, or if reinserted due to nausea and vomiting after removal by POD 3 and the patient is unable to tolerate a solid diet on POD 7, but starts a solid diet before POD 14.
  Grade B DGE: If the NGT is needed from POD 8-14, if reinserted after POD 7, or if the patient cannot tolerate unlimited oral intake by POD 14, but is able to resume a solid diet before POD 21.
  Grade C DGE: When nasogastric intubation cannot be discontinued or has to be reinserted after POD 14, or if the patient is unable to maintain unlimited oral intake by POD 21.
  PS- Higher the score worst the outcome.
Morbidity- Postoperative pancreatic fistula (POPF) | 30days following the pancreaticoduodenectomy
  A POPF is an abnormal communication between the pancreatic ductal epithelium and another epithelial surface containing pancreas-derived enzyme-rich fluid.
  Biochemical leak (Grade A): Pancreatic fistula often appears well and requires no intervention.
  Grade B: Pancreatic fistulas occur in patients who generally appear well, but may require parenteral nutrition or interventional fistula drainage for the fistula to heal.
  Grade C: Pancreatic fistulas, in which patients appear ill and require parenteral nutrition, interventional drainage, and potentially even re-operation for treatment.
  PS- Higher the score worst the outcome.
Morbidity- Post pancreatectomy Hemorrhage (PPH) | 30days following the pancreaticoduodenectomy
  Time of onset
  * Early hemorrhage ( 24 h after the end of the index operation)
  * Late hemorrhage ( 24 h after the end of the index operation)
  Location
  * Intraluminal
  * Extraluminal
  Severity of Hemorrhage Mild
  * Small or medium volume blood loss (from drains, nasogastric tube, or on ultrasonography, decrease in hemoglobin concentration 3 g/dl)
  * Mild clinical impairment of the patient, no therapeutic consequence, or at most the need for noninvasive treatment with volume resuscitation or blood transfusions (2-3 units packed cells within 24hrs of end of operation or 1-3 units if later than 24hrs after operation)
  * No need for reoperation or interventional angiographic embolization; endoscopic treatment of anastomotic bleeding may occur provided the other conditions apply
  Severe
  * Large volume blood loss (drop in hemoglobin level by 3g/dl)
  * Clinically significant impairment and need for blood transfusion (3 units packed cells)
  * Need for invasive treatment.
Mortality | 30days following the pancreaticoduodenectomy
  Survival within 30days.

CONTACTS AND LOCATIONS:
Overall Officials: Harish Neupane, MBBS, MS, Study Chair — Chitwan Medical Hospital
Locations (1):
- Chitwan Medical College Teaching Hospital, Bharatpur, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: Undecided
IPD can be shared in view of the progress of medical research. An interested person should contact the primary investigator.

REFERENCES:
- [Background] Ruiz-Tovar J, Martin-Perez E, Fernandez-Contreras ME, Reguero-Callejas ME, Gamallo-Amat C. Impact of preoperative levels of hemoglobin and albumin on the survival of pancreatic carcinoma. Rev Esp Enferm Dig. 2010 Nov;102(11):631-6. doi: 10.4321/s1130-01082010001100003. PMID 21142383
- [Background] Shirai Y, Shiba H, Haruki K, Horiuchi T, Saito N, Fujiwara Y, Sakamoto T, Uwagawa T, Yanaga K. Preoperative Platelet-to-Albumin Ratio Predicts Prognosis of Patients with Pancreatic Ductal Adenocarcinoma After Pancreatic Resection. Anticancer Res. 2017 Feb;37(2):787-793. doi: 10.21873/anticanres.11378. PMID 28179331
- [Background] Xu SS, Li S, Xu HX, Li H, Wu CT, Wang WQ, Gao HL, Jiang W, Zhang WH, Li TJ, Ni QX, Liu L, Yu XJ. Haemoglobin, albumin, lymphocyte and platelet predicts postoperative survival in pancreatic cancer. World J Gastroenterol. 2020 Feb 28;26(8):828-838. doi: 10.3748/wjg.v26.i8.828. PMID 32148380
- [Background] Gao X, Lin B, Lin Q, Ye T, Zhou T, Hu M, Zhu H, Lu F, Chen W, Xia P, Zhang F, Yu Z. A HALP score-based prediction model for survival of patients with the upper tract urothelial carcinoma undergoing radical nephroureterectomy. Bosn J Basic Med Sci. 2022 Apr 1;22(2):280-290. doi: 10.17305/bjbms.2021.6543. PMID 35020581
- [Background] Guo Y, Shi D, Zhang J, Mao S, Wang L, Zhang W, Zhang Z, Jin L, Yang B, Ye L, Yao X. The Hemoglobin, Albumin, Lymphocyte, and Platelet (HALP) Score is a Novel Significant Prognostic Factor for Patients with Metastatic Prostate Cancer Undergoing Cytoreductive Radical Prostatectomy. J Cancer. 2019 Jan 1;10(1):81-91. doi: 10.7150/jca.27210. eCollection 2019. PMID 30662528
- [Background] Wang X, He Q, Liang H, Liu J, Xu X, Jiang K, Zhang J. A novel robust nomogram based on preoperative hemoglobin and albumin levels and lymphocyte and platelet counts (HALP) for predicting lymph node metastasis of gastric cancer. J Gastrointest Oncol. 2021 Dec;12(6):2706-2718. doi: 10.21037/jgo-21-507. PMID 35070400
- [Background] Leetanaporn K, Hanprasertpong J. Predictive Value of the Hemoglobin-Albumin-Lymphocyte-Platelet (HALP) Index on the Oncological Outcomes of Locally Advanced Cervical Cancer Patients. Cancer Manag Res. 2022 Jun 14;14:1961-1972. doi: 10.2147/CMAR.S365612. eCollection 2022. PMID 35726336
- [Background] Bassi C, Marchegiani G, Dervenis C, Sarr M, Abu Hilal M, Adham M, Allen P, Andersson R, Asbun HJ, Besselink MG, Conlon K, Del Chiaro M, Falconi M, Fernandez-Cruz L, Fernandez-Del Castillo C, Fingerhut A, Friess H, Gouma DJ, Hackert T, Izbicki J, Lillemoe KD, Neoptolemos JP, Olah A, Schulick R, Shrikhande SV, Takada T, Takaori K, Traverso W, Vollmer CM, Wolfgang CL, Yeo CJ, Salvia R, Buchler M; International Study Group on Pancreatic Surgery (ISGPS). The 2016 update of the International Study Group (ISGPS) definition and grading of postoperative pancreatic fistula: 11 Years After. Surgery. 2017 Mar;161(3):584-591. doi: 10.1016/j.surg.2016.11.014. Epub 2016 Dec 28. PMID 28040257
- [Background] Wente MN, Veit JA, Bassi C, Dervenis C, Fingerhut A, Gouma DJ, Izbicki JR, Neoptolemos JP, Padbury RT, Sarr MG, Yeo CJ, Buchler MW. Postpancreatectomy hemorrhage (PPH): an International Study Group of Pancreatic Surgery (ISGPS) definition. Surgery. 2007 Jul;142(1):20-5. doi: 10.1016/j.surg.2007.02.001. PMID 17629996
- [Background] Wente MN, Bassi C, Dervenis C, Fingerhut A, Gouma DJ, Izbicki JR, Neoptolemos JP, Padbury RT, Sarr MG, Traverso LW, Yeo CJ, Buchler MW. Delayed gastric emptying (DGE) after pancreatic surgery: a suggested definition by the International Study Group of Pancreatic Surgery (ISGPS). Surgery. 2007 Nov;142(5):761-8. doi: 10.1016/j.surg.2007.05.005. PMID 17981197
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912
- [Result] Hoshimoto S, Hishinuma S, Shirakawa H, Tomikawa M, Ozawa I, Ogata Y. Validation and clinical usefulness of pre- and postoperative systemic inflammatory parameters as prognostic markers in patients with potentially resectable pancreatic cancer. Pancreatology. 2020 Mar;20(2):239-246. doi: 10.1016/j.pan.2019.12.004. Epub 2019 Dec 14. PMID 31862230
- [Result] Afaneh C, Gerszberg D, Slattery E, Seres DS, Chabot JA, Kluger MD. Pancreatic cancer surgery and nutrition management: a review of the current literature. Hepatobiliary Surg Nutr. 2015 Feb;4(1):59-71. doi: 10.3978/j.issn.2304-3881.2014.08.07. PMID 25713805